CLINICAL TRIAL: NCT00574639
Title: Mechanisms of Hypoglycemia-Associated Autonomic Dysfunction. The Effect of Alprazolam on Exercise Induced Hypoglycemia.
Brief Title: Mechanisms of Hypoglycemia Associated Autonomic Dysfunction Question 2
Acronym: Alp Ex
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00044868; HL056693
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Alprazolam; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — Alprazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): Day 1 study two hyperinsulinemic (high Insulin dose) euglycemic (normal glucose level) clamps x 2. Day 2 exercise for 90 minutes on recumbent bike. Patient randomized to placebo or Xanax (Alprazolam) drug on Day 1 to receive 1 mg orally prior to each clamp.
  Interventions: Drug: Alprazolam
- Arm 2 (Experimental): Day 1 study two hyperinsulinemic (high Insulin dose) euglycemic (normal glucose level) clamps x 2. Day 2 exercise for 90 minutes on recumbent bike. Patient randomized to placebo or Xanax (Alprazolam) drug on Day 1 to receive 1 mg orally prior to each clamp.
  Interventions: Drug: Placebo
- Arm 3 (Experimental): Day 1 study two hyperinsulinemic (high Insulin dose) hypoglycemic (low glucose level) clamps x 2. Day 2 exercise for 90 minutes on recumbent bike. Patient randomized to placebo or Xanax (Alprazolam) drug on Day 1 to receive 1 mg orally prior to each clamp.
  Interventions: Drug: Alprazolam
- Arm 4 (Experimental): Day 1 study two hyperinsulinemic (high Insulin dose) hypoglycemic (low glucose level) clamps x 2. Day 2 exercise for 90 minutes on recumbent bike. Patient randomized to placebo or Xanax (Alprazolam) drug on Day 1 to receive 1 mg orally prior to each clamp.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alprazolam — 1 mg given orally prior to morning and afternoon clamps on Day 1
  Other Names: Xanax
  Arms: Arm 1; Arm 3
Drug: Placebo — 1 mg given orally prior to glucose clamps on Day 1 (morning and afternoon)
  Arms: Arm 2; Arm 4

SUMMARY:
The purpose of this study is to determine the way by which Alprazolam (Xanax) an anti-anxiety drug affects specialized molecules in your brain called GABA (A) receptors that alter your body's ability to defend itself from low blood sugar (hypoglycemia). We hypothesize that prior activation of GABA (A) receptors may result in blunting of counterregulatory responses during subsequent hypoglycemia and exercise.

DETAILED DESCRIPTION:
The ultimate goal of this project is to identify treatments and approaches that will allow patients with diabetes to enjoy all the benefits of good glycemic control without the damaging limitations of severe hypoglycemia. The specific aim of this study is to determine if gamma aminobutyric acid (GABA A) receptors plays a role in the development of exercise associated autonomic dysfunction in type 1 diabetes and healthy man.

ELIGIBILITY:
Inclusion

* 14 Type 1 DM patients (7 male and 7 female) aged 18-50 years
* HBA1c > 6%
* BMI<35 kg/m2
* 14 healthy individuals (7 male and 7 female) aged 18-50 years, BMI matched

Exclusion

* Pregnant women
* Subjects unable to give voluntary informed consent
* Subjects on anticoagulant drugs, anemic or with known bleeding diatheses
* Subjects taking any of the following medications will be excluded: Non-selective Beta Blockers, Sedative-Hypnotics, Anticonvulsants, Antiparkinsonian drugs, Antipsychotics, Antidepressants, Mood stabilizers, CNS Stimulants, Opioids, Hallucinogens
* Subjects with a recent medical illness
* Subjects with a history of hypertension, heart disease, cerebrovascular incidents
* Subjects with known liver or kidney disease Physical Exam Exclusion Criteria
* History of uncontrolled severe hypertension (i.e., blood pressure greater than 150/95)
* Clinically significant Cardiac Abnormalities (e.g. Heart Failure, Arrhythmia)
* Pneumonia
* Hepatic Failure /Jaundice
* Renal Failure
* Acute Cerebrovascular/ Neurological deficit
* Fever greater than 38.0 C

Screening Laboratory blood tests Exclusion Criteria according to protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Epinephrine Levels | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Hedrington MS, Tate DB, Younk LM, Davis SN. Effects of Antecedent GABA A Receptor Activation on Counterregulatory Responses to Exercise in Healthy Man. Diabetes. 2015 Sep;64(9):3253-61. doi: 10.2337/db15-0212. Epub 2015 Apr 21. PMID 25901095